CLINICAL TRIAL: NCT00573170
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, Crossover Study to Evaluate the Efficacy of TREXIMET® (Sumatriptan + Naproxen Sodium) vs. Butalbital-containing Combination Medications for the Acute Treatment of Migraine When Administered During the Moderate-Severe Migraine Pain, Studies 1 and 2 of 2
Brief Title: TREXIMET® Versus Butalbital-containing Combination Medications for the Acute Treatment of Migraine in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TRX109011/TRX109013; NCT00599157 (obsolete NCT alias); NCT01812408 (obsolete NCT alias)
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Results first posted 2010-12-29 (Estimated); Last update posted 2010-12-29 (Estimated); Status verified 2010-11

CONDITIONS: Migraine Disorders; Migraine, Acute
Keywords: Migraine, acute; Migraine; Butalbital-containing Combination Medication (BCM); Naproxen sodium; Sumatriptan succinate; TREXIMET®
MeSH Terms: conditions — Migraine Disorders | interventions — sumatriptan-naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- TPB (Other): TREXIMET® (Attack 1), placebo (Attack 2), BCM (Attack 3)
  Interventions: Drug: TREXIMET®; Drug: Butalbital-containing Combination Medications (BCM); Drug: placebo
- TBP (Other): TREXIMET® (Attack 1), BCM (Attack 2), placebo (Attack 3)
  Interventions: Drug: TREXIMET®; Drug: Butalbital-containing Combination Medications (BCM); Drug: placebo
- BTP (Other): BCM (Attack 1), TREXIMET® (Attack 2), placebo (Attack 3)
  Interventions: Drug: TREXIMET®; Drug: Butalbital-containing Combination Medications (BCM); Drug: placebo
- BPT (Other): BCM (Attack 1), placebo (Attack 2), TREXIMET® (Attack 3)
  Interventions: Drug: TREXIMET®; Drug: Butalbital-containing Combination Medications (BCM); Drug: placebo
- PTB (Other): placebo (Attack 1), TREXIMET® (Attack 2), BCM (Attack 3)
  Interventions: Drug: TREXIMET®; Drug: Butalbital-containing Combination Medications (BCM); Drug: placebo
- PBT (Other): placebo (Attack 1), BCM (Attack 2), TREXIMET® (Attack 3)
  Interventions: Drug: TREXIMET®; Drug: Butalbital-containing Combination Medications (BCM); Drug: placebo

INTERVENTIONS:
Drug: TREXIMET® — Sumatriptan + Naproxen Sodium (fixed dose combination tablet of sumatriptan succinate [equivalent to sumatriptan 85mg] and naproxen sodium 500mg)
Drug: Butalbital-containing Combination Medications (BCM) — butalbital-containing combination medication (BCM; acetaminophen 325mg, caffeine 40mg, and butalbital 50mg) [currently marketed as Fioricet]
Drug: placebo — placebo

SUMMARY:
Study TRX109011/TRX109013, A Randomized, Double-blind, Double-dummy, Placebo-controlled, Crossover Study to Evaluate the Efficacy of TREXIMET® (Sumatriptan + Naproxen Sodium) versus Butalbital-containing Combination Medications (BCM) for the Acute Treatment of Migraine when administered during the Moderate-Severe Pain Phase of the Migraine (Studies 1 and 2 of 2)

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, double-dummy, placebo-controlled, crossover, three-attack, outpatient study in which TREXIMET® will be compared to a butalbital-containing combination medication (BCM; acetaminophen 325mg, caffeine 40mg, and butalbital 50mg [Fioricet]) for the acute treatment of migraine headaches. Subjects will be randomized to one of 6 possible treatment sequences (TPB, TBP, BTP, BPT, PTB, PBT where T = TREXIMET®; P = Placebo; B = Butalbital-containing Combination Medication) . Subjects will treat each of the 3 migraine attacks when pain is moderate to severe. The study will include 4 visits: (1) a Screening visit at study entry, (2) a Drug Screen visit, (3) a Randomization visit, and (4) a Final visit. The Final visit occurs either (A) upon withdrawal or (B) after treatment of 3 migraine attacks. The primary objective is to evaluate the efficacy of TREXIMET® versus BCM for the acute treatment of moderate/severe migraine. These two replicate studies were amended while ongoing to allow for the reporting of pooled data only.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 65 years. Female subjects are eligible for participation if they are either of non-childbearing potential (not capable of becoming pregnant) OR of childbearing potential having a negative urine pregnancy test at screening, and using contraception if sexually active. If using oral contraceptives, the subjects should be on a stable regimen of oral contraceptives (>/= 2 months).

Eligible subjects must:

* have migraine with or without aura (2004 ICHD-II criteria) and must have had at least 2 attacks per month meeting these criteria in the three months prior to screening.
* have documented use of Butalbital-containing Combination Medication (MCM) to have treated at least one migraine.
* be able to understand how to complete the cognitive assessments and all other questionnaires programmed in an electronic diary.
* be willing and able to provide written informed consent.

Exclusion Criteria:

A subject is not eligible if they have:

* >8 migraines or >/= 15 headache days per month in total, or has retinal, basilar, or hemiplegic migraine, or secondary headaches.
* taken >350mg/day of butalbital and/or other barbiturates on an equivalent dose basis, on average, over the 30 days prior to screening.
* is likely to have unrecognized cardiovascular or cerebrovascular disease (based on history or risk factors).
* blood pressure >/= 140/90mmHg in 2 out of 3 BP measurements or is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker.
* history of congenital heart disease, cardiac arrhythmias requiring medication, or a clinical significant electrocardiogram abnormality.
* evidence or history of any ischemic vascular disease including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or signs/symptoms consistent with these.
* evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower the convulsive threshold; or has been treated with an antiepileptic drug for seizure control within 5 years prior to screening.
* a history of impaired hepatic or renal function that contraindicates participation in the study.
* hypersensitivity, allergy, intolerance, or contraindication to the use of any triptan, NSAID, aspirin, barbiturates, or acetaminophen (including all sumatriptan and naproxen preparations), has porphyria or has nasal polyps and asthma.
* is currently taking, or has taken in the previous three months, an ergot preparation for migraine prophylaxis; or is taking a migraine or prophylactic medication that is not stabilized (i.e. a change of dose within the last 2 months) for either chronic or intermittent migraine prophylaxis or for a co-morbid condition that is not stabilized.
* a recent history of regular use of opioids (including opioids in combination with butalbital, e.g. Fioricet with codeine) or barbiturates other than butalbital. Regular use is defined as an average of 4 days per month over the last 6 months.
* taken, or plans to take, a monoamine oxidase inhibitor (MAOI), including herbal preparations containing St. John's Wort (Hypericum perforatum), anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
* history of any bleeding disorder or is currently taking any anti-coagulant or any antiplatelet agent (except low-dose aspirin </= 325mg/day for cardioprotective reasons).
* evidence or history of any gastrointestinal surgery or GI ulceration or perforation in the past six months, gastrointestinal bleeding in the past year; or evidence or history of inflammatory bowel disease.
* is pregnant, actively trying to become pregnant, breast feeding, or not willing to have pregnancy test performed.
* evidence of alcohol or substance abuse within the last year or any concurrent medical or psychiatric condition which, in the investigator's judgement, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical study.
* participated in an investigational drug trial within the previous four weeks or plans to participate in another study at any time during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (98):
- United States (98):
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tempe, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSk Investigational Site, Anaheim, California
  - GSK Investigational Site, Garden Grove, California
  - GSK Investigational Site, Irvine, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Sherman Oaks, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Westlake Village, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, East Hartford, Connecticut
  - GSK Investigational Site, New Britain, Connecticut
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Naples, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Rome, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Gurnee, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Paducah, Kentucky
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Biddeford, Maine
  - GSK Investigational Site, Pikesville, Maryland
  - GSk Investigational Site, Brockton, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Hattiesburg, Mississippi
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Ridgewood, New Jersey
  - GSK Investigational Site, Stratford, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Mount Vernon, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Orchard Park, New York
  - GSK Investigational Site, Schenectady, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Valley Stream, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Bismarck, North Dakota
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Minot, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Greensburg, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Warwick, Rhode Island
  - GSK Investigational Site, Beaufort, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSk Investigational Site, Rapid City, South Dakota
  - GSK Investigational Site, Columbia, Tennessee
  - GSK Investigational Site, Cordova, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Virginia Beach, Virginia

REFERENCES:
- [Background] Silberstein SD, McCrory DC. Butalbital in the treatment of headache: history, pharmacology, and efficacy. Headache. 2001 Nov-Dec;41(10):953-67. doi: 10.1046/j.1526-4610.2001.01189.x. PMID 11903523
- [Background] Bigal ME, Rapoport AM, Sheftell FD, Tepper SJ, Lipton RB. Transformed migraine and medication overuse in a tertiary headache centre--clinical characteristics and treatment outcomes. Cephalalgia. 2004 Jun;24(6):483-90. doi: 10.1111/j.1468-2982.2004.00691.x. PMID 15154858
- [Background] Wenzel RG, Sarvis CA. Do butalbital-containing products have a role in the management of migraine? Pharmacotherapy. 2002 Aug;22(8):1029-35. doi: 10.1592/phco.22.12.1029.33595. PMID 12173787
- [Derived] Derosier F, Sheftell F, Silberstein S, Cady R, Ruoff G, Krishen A, Peykamian M. Sumatriptan-naproxen and butalbital: a double-blind, placebo-controlled crossover study. Headache. 2012 Apr;52(4):530-43. doi: 10.1111/j.1526-4610.2011.02039.x. Epub 2011 Nov 21. PMID 22103635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Results for the TRX109011 (NCT00573170) and TRX109013 (NCT00599157) studies were pooled for analysis. Individual studies were not analyzed or reported separately. The individual protocols were amended while ongoing to allow for pooling of study data for analysis.
Pre-assignment Details: Randomized participants were treated for three separate migraine attacks with three different investigational products, assigned in randomized order, as one of six possible treatment sequences. Not all participants enrolled in the study were randomized for treatment; those participants who were randomized are said to have "started" the study
Groups:
- Treximet, Placebo, Butalbital-containing Combo. Medication: Fixed dose combination (combo.) tablet of sumatriptan succinate (equivalent to sumatriptan 85 milligrams [mg]) and naproxen sodium 500 mg (Treximet) for treatment of first migraine attack, followed by a 7-day washout period; matching placebo for treatment of second migraine attack, followed by a 7-day washout period; comparator of acetaminophen 325 mg, caffeine 40 mg, and butalbital 50 mg (butalbital-containing combination medication), currently marketed as Fioricet, for treatment of third migraine attack. Treatment of each separate migraine attack had to be preceeded by a 24-hour pain-free period to ensure that a separate migraine attack was being treated.
- Treximet, Butalbital-containing Combo. Medication, Placebo: Fixed dose combination tablet of sumatriptan succinate (equivalent to sumatriptan 85 milligrams [mg]) and naproxen sodium 500 mg (Treximet) for treatment of first migraine attack, followed by a 7-day washout period; comparator of acetaminophen 325 mg, caffeine 40 mg, and butalbital 50 mg (butalbital-containing combination medication), currently marketed as Fioricet, for treatment of second migraine attack, followed by a 7-day washout period; matching placebo for treatment of third migraine attack, followed by a 7-day washout period. Treatment of each separate migraine attack had to be preceeded by a 24-hour pain-free period to ensure that a separate migraine attack was being treated.
- Butalbital-containing Combo. Medication, Treximet, Placebo: Comparator of acetaminophen 325 mg, caffeine 40 mg, and butalbital 50 mg (butalbital-containing combination medication), currently marketed as Fioricet, for treatment of first migraine attack, followed by a 7-day washout period; fixed dose combination tablet of sumatriptan succinate (equivalent to sumatriptan 85 milligrams [mg]) and naproxen sodium 500 mg (Treximet) for treatment of second migraine attack, followed by a 7-day washout period; matching placebo for treatment of third migraine attack, followed by a 7-day washout period. Treatment of each separate migraine attack had to be preceeded by a 24-hour pain-free period to ensure that a separate migraine attack was being treated.
- Butalbital-containing Combo. Medication, Placebo, Treximet: Comparator of acetaminophen 325 mg, caffeine 40 mg, and butalbital 50 mg (butalbital-containing combination medication), currently marketed as Fioricet, for treatment of first migraine attack, followed by a 7-day washout period; matching placebo for treatment of second migraine attack, followed by a 7-day washout period; fixed dose combination tablet of sumatriptan succinate (equivalent to sumatriptan 85 milligrams [mg]) and naproxen sodium 500 mg (Treximet) for treatment of third migraine attack. Treatment of each separate migraine attack had to be preceeded by a 24-hour pain-free period to ensure that a separate migraine attack was being treated.
- Placebo, Treximet, Butalbital-containing Combo. Medication: Matching placebo for treatment of first migraine attack, followed by a 7-day washout period; fixed dose combination tablet of sumatriptan succinate (equivalent to sumatriptan 85 milligrams [mg]) and naproxen sodium 500 mg (Treximet) for treatment of second migraine attack, followed by a 7-day washout period; comparator of acetaminophen 325 mg, caffeine 40 mg, and butalbital 50 mg (butalbital-containing combination medication), currently marketed as Fioricet, for treatment of third migraine attack. Treatment of each separate migraine attack had to be preceeded by a 24-hour pain-free period to ensure that a separate migraine attack was being treated.
- Placebo, Butalbital-containing Combo. Medication, Treximet: Matching placebo for treatment of first migraine attack, followed by a 7-day washout period; comparator of acetaminophen 325 mg, caffeine 40 mg, and butalbital 50 mg (butalbital-containing combination medication), currently marketed as Fioricet, for treatment of second migraine attack, followed by a 7-day washout period; fixed dose combination tablet of sumatriptan succinate (equivalent to sumatriptan 85 milligrams [mg]) and naproxen sodium 500 mg (Treximet) for treatment of third migraine attack. Treatment of each separate migraine attack had to be preceeded by a 24-hour pain-free period to ensure that a separate migraine attack was being treated.
Period: First Treatment Period
Arm/Group | Treximet, Placebo, Butalbital-containing Combo. Medication | Treximet, Butalbital-containing Combo. Medication, Placebo | Butalbital-containing Combo. Medication, Treximet, Placebo | Butalbital-containing Combo. Medication, Placebo, Treximet | Placebo, Treximet, Butalbital-containing Combo. Medication | Placebo, Butalbital-containing Combo. Medication, Treximet
Started | 64 | 60 | 60 | 66 | 63 | 62
Completed | 64 | 60 | 60 | 66 | 62 | 62
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Did Not Treat Attack 1 | 0 | 0 | 0 | 0 | 1 | 0
Period: First Washout Period
Arm/Group | Treximet, Placebo, Butalbital-containing Combo. Medication | Treximet, Butalbital-containing Combo. Medication, Placebo | Butalbital-containing Combo. Medication, Treximet, Placebo | Butalbital-containing Combo. Medication, Placebo, Treximet | Placebo, Treximet, Butalbital-containing Combo. Medication | Placebo, Butalbital-containing Combo. Medication, Treximet
Started | 64 | 60 | 60 | 66 | 62 | 62
Completed | 56 | 58 | 59 | 61 | 59 (Source data list 4 noncompleters; per number starting next period, there were only 3 noncompleters.) | 55
Not Completed | 8 | 2 | 1 | 5 | 3 | 7
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 3 | 3
Not completed — Other | 4 | 0 | 1 | 1 | 0 | 0
Period: Second Treatment Period
Arm/Group | Treximet, Placebo, Butalbital-containing Combo. Medication | Treximet, Butalbital-containing Combo. Medication, Placebo | Butalbital-containing Combo. Medication, Treximet, Placebo | Butalbital-containing Combo. Medication, Placebo, Treximet | Placebo, Treximet, Butalbital-containing Combo. Medication | Placebo, Butalbital-containing Combo. Medication, Treximet
Started | 56 | 58 | 59 | 61 | 59 | 55
Completed | 56 | 58 | 59 | 61 | 59 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Washout Period
Arm/Group | Treximet, Placebo, Butalbital-containing Combo. Medication | Treximet, Butalbital-containing Combo. Medication, Placebo | Butalbital-containing Combo. Medication, Treximet, Placebo | Butalbital-containing Combo. Medication, Placebo, Treximet | Placebo, Treximet, Butalbital-containing Combo. Medication | Placebo, Butalbital-containing Combo. Medication, Treximet
Started | 56 | 58 | 59 | 61 | 59 | 55
Completed | 51 | 54 | 55 | 56 | 51 | 53
Not Completed | 5 | 4 | 4 | 5 | 8 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other | 1 | 2 | 1 | 4 | 6 | 2
Period: Third Treatment Period
Arm/Group | Treximet, Placebo, Butalbital-containing Combo. Medication | Treximet, Butalbital-containing Combo. Medication, Placebo | Butalbital-containing Combo. Medication, Treximet, Placebo | Butalbital-containing Combo. Medication, Placebo, Treximet | Placebo, Treximet, Butalbital-containing Combo. Medication | Placebo, Butalbital-containing Combo. Medication, Treximet
Started | 51 | 54 | 55 | 56 | 51 | 53
Completed | 50 | 54 | 55 | 56 | 51 | 51
Not Completed | 1 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants Treated at Least Once: All study participants who were treated at least once with study medication
Arm/Group | All Study Participants Treated at Least Once
Number analyzed (Participants) | 442
Age Continuous [Mean (Standard Deviation); unit: Years] — Baseline data are reported for the Safety Population, comprised of all participants who were treated at least once with study medication. . All randomized participants are accounted for in the Participant Flow module. Only a portion of the participants who were randomized comprise the Safety Population.
  Years | 42.6 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 391
  Male | 51
Race/Ethnicity, Customized [Number; unit: participants]
  White-White/Caucasian/European Heritage | 368
  African American/African Heritage | 61
  Mixed Race | 4
  Asian - Central/South | 2
  Asian - South East Asian Heritage | 2
  White - Arabic/North African Heritage | 2
  American Indian or Native Alaskan | 1
  Asian - Japanese Heritage | 1
  Native Hawaiian or Other Pacific Islander | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Sustained Pain-free (SPF) Response From 2 to 24 Hours Post-dose
Description: SPF 2-24 hours is defined for all participants as having no pain at 2 hours post-dose and without the return of any pain or the use of any rescue medication (any medication taken after the first dose of study medication for any migraine pain or symptoms) from 2-24 hours.
Time Frame: From 2 to 24 hours post-dose. All 3 migraine attacks were to have been treated within 19 weeks of randomization (when study medication was dispensed).
Population: Intent-to-Treat (ITT) Population: all participants who were treated with investigational product and provided at least one post-dose efficacy assessment . Participants may have been included in one, two, or all of the Placebo, Treximet and Butalbital-containing combination medication arms due to the cross-over nature of the study design.
Measure: Number; unit: participants
Groups:
- Placebo: Attacks for which treatment of moderate or severe pain was placebo
- Treximet: Attacks for which treatment of moderate or severe pain was Treximet
- Butalbital-containing Combination Medication: Attacks for which treatment of moderate or severe pain was Butalbital-containing combination medication
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 320 | 317 | 304
participants | 10 | 26 | 18
Statistical Analysis 1: Comparison: Treximet vs Butalbital-containing Combination Medication; Test type: Superiority or Other; p = 0.378, Generalized Estimating Equations — Compares odds ratio; Odds Ratio (OR) = 1.3, 95% CI 2-sided [0.7 to 2.5]

2. Secondary Outcome: Number of Participants With a Pain-free Response From 2 to 48 Hours Post-dose
Description: Pain-Free is defined as having no pain and without the use of any rescue medication from the time of the initial dose of study medication for a particular migraine attack until the defined time point at 2, 4, 6, 8, 24 or 48 hours post-dose.
Time Frame: At 2, 4, 6, 8, 24, and 48 hours post-dose for each attack treated with study medication. All 3 migraine attacks were to have been treated within 19 weeks of randomization (when study medication was dispensed).
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 320 | 317 | 304
participants
  2 hours post-dose | 16 | 45 | 26
  4 hours post-dose | 21 | 86 | 39
  6 hours post-dose | 29 | 78 | 40
  8 hours post-dose | 30 | 79 | 42
  24 hours post-dose | 48 | 104 | 78
  48 hours post-dose | 51 | 93 | 66

3. Secondary Outcome: Number of Participants Using Rescue Medication Within 48 Hours Post Dose
Description: Number of participants who took any medication to treat their migraine pain or symptoms within 48 hours after they took the first dose of study medication (placebo, Treximet, or butalbital-containing combination medication) for that attack. Participants were asked not to take rescue for at least 2 hours after they took the study medication (placebo, Treximet, or butalbital-containing combination medication) for that attack. Participants took rescue medication if they felt they needed it.
Time Frame: From dose time through 48 hours post-dose for each attack treated with study medication. All 3 migraine attacks were to have been treated within 19 weeks of randomization (when study medication was dispensed).
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 320 | 317 | 304
participants
  Use of 1st rescue < 2 hours post-dose | 25 | 19 | 25
  Use of 1st rescue (investigational medication) | 234 | 158 | 203
  Use of 2nd rescue (investigational medication) | 114 | 79 | 121
  Use of other rescue (not investigational med.) | 6 | 5 | 8

4. Secondary Outcome: Mean Time to First Use of Rescue Medication for the First Attack Treated With Study Medication (Attack 1)
Description: Average time until participants took any medication to treat their migraine pain or symptoms within 48 hours after they took the first dose of study medication (placebo, Treximet, or butalbital-containing combination medication) for the first migraine attack treated. Participants were asked not to take rescue for at least 2 hours after they took the study medication (placebo, Treximet, or butalbital-containing combination medication) for that attack. Participants took rescue medication if they felt they needed it.
Time Frame: as for outcome 3
Population: Participants in the ITT population who treated migraine Attack 1 with study medication and then used migraine rescue medication after dosing.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Placebo: Participants taking any rescue medication within 48 hours of treating Migraine Attack 1 with placebo
- Treximet: Participants taking any rescue medication within 48 hours of treating Migraine Attack 1 with Treximet
- Butalbital-containing Combination Medication: Participants taking any rescue medication within 48 hours of treating Migraine Attack 1 with Butalbital-containing combination medication
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 74 | 52 | 67
hours | 12.00 (1.44) | 17.07 (1.22) | 20.15 (2.07)

5. Secondary Outcome: Mean Time to First Use of Rescue Medication for the Second Attack Treated With Study Medication (Attack 2)
Description: Average time until participants took any medication to treat their migraine pain or symptoms within 48 hours after they took the first dose of study medication (placebo, Treximet, or butalbital-containing combination medication) for their second migraine attack treated in the study. Participants were asked not to take rescue for at least 2 hours after they took the study medication (placebo, Treximet, or butalbital-containing combination medication) for that attack. Participants took rescue medication if they felt they needed it.
Time Frame: as for outcome 3
Population: Participants in the ITT population who treated migraine Attack 2 with study medication and then used migraine rescue medication after dosing.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Placebo: Participants taking any rescue medication within 48 hours of treating Migraine Attack 2 with placebo
- Treximet: Participants taking any rescue medication within 48 hours of treating Migraine Attack 2 with Treximet
- Butalbital-containing Combination Medication: Participants taking any rescue medication within 48 hours of treating Migraine Attack 2 with Butalbital-containing combination medication
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 90 | 55 | 72
hours | 8.29 (1.12) | 20.90 (1.64) | 16.70 (2.05)

6. Secondary Outcome: Mean Time to First Use of Rescue Medication for the Third Attack Treated With Study Medication (Attack 3)
Description: Average time until participants took any medication to treat their migraine pain or symptoms within 48 hours after they took the first dose of study medication (placebo, Treximet, or butalbital-containing combination medication) for their third migraine attack treated in the study. Participants were asked not to take rescue for at least 2 hours after they took the study medication (placebo, Treximet, or butalbital-containing combination medication) for that attack. Participants took rescue medication if they felt they needed it.
Time Frame: as for outcome 3
Population: Participants in the ITT population who treated migraine Attack 3 with study medication and then used migraine rescue medication after dosing.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Placebo: Participants taking any rescue medication within 48 hours of treating Migraine Attack 3 with placebo
- Treximet: Participants taking any rescue medication within 48 hours of treating Migraine Attack 3 with Treximet
- Butalbital-containing Combination Medication: Participants taking any rescue medication within 48 hours of treating Migraine Attack 3 with Butalbital-containing combination medication
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 72 | 58 | 65
hours | 6.69 (0.58) | 20.77 (1.93) | 9.44 (1.10)

7. Secondary Outcome: Number of Participants With a Migraine-free Response 2-48 Hours After Dosing
Description: Migraine-free is defined as pain-free with no migraine-associated symptoms (nausea, vomiting, photophobia [sensitivity to light], and phonophobia [sensitivity to sound]) with use of any rescue medication before the defined time point.
Time Frame: as for outcome 2
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 320 | 317 | 304
participants
  2 hours | 14 | 33 | 22
  4 hours | 20 | 74 | 37
  6 hours | 28 | 70 | 39
  8 hours | 29 | 73 | 40
  24 hours | 46 | 101 | 75
  48 hours | 48 | 90 | 65

8. Secondary Outcome: Number of Participants With Pain-freedom and Relief of Nausea at 2, 4, 6, 8, 24 and 48 Post-dose Time Points
Description: The number of participants with no pain and relief of nausea in those participants for whom nausea was present at dose time. Participants using rescue medication were removed from the participants with relief group for all subsequent timed assessments, regardless of pain and associated symptom evaluations at the specified time point.
Time Frame: as for outcome 2
Population: ITT Population - including only those participants who reported nausea at dose time.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 152 | 154 | 133
participants
  2 hrs post-dose | 5 | 13 | 8
  4 hrs post-dose | 6 | 28 | 8
  6 hrs post-dose | 8 | 32 | 8
  8 hrs post-dose | 9 | 29 | 9
  24 hrs post-dose | 15 | 39 | 30
  48 hrs post-dose | 20 | 41 | 28

9. Secondary Outcome: Number of Participants With Pain-freedom and Relief of Photophobia at 2, 4, 6, 8, 24 and 48 Post-dose Time Points
Description: The number of participants with no pain and relief of photophobia in those participants for whom photophobia was present at dose time. Participants using rescue medication were removed from the participants with relief group for all subsequent timed assessments, regardless of pain and associated symptom evaluations at the specified time point.
Time Frame: as for outcome 2
Population: ITT Population - including only those participants who reported photophobia at dose time.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 277 | 269 | 251
participants
  2 hrs post-dose | 11 | 30 | 16
  4 hrs post-dose | 16 | 64 | 23
  6 hrs post-dose | 22 | 54 | 27
  8 hrs post-dose | 21 | 61 | 32
  24 hrs post-dose | 35 | 84 | 24
  48 hrs post-dose | 38 | 81 | 20

10. Secondary Outcome: Number of Participants With Pain-freedom and Relief of Phonophobia at 2, 4, 6, 8, 24 and 48 Post-dose Time Points
Description: The number of participants with no pain and relief of phonophobia in those participants for whom phonophobia was present at dose time. Participants using rescue medication were removed from the participants with relief group for all subsequent timed assessments, regardless of pain and associated symptom evaluations at the specified time point.
Time Frame: as for outcome 2
Population: ITT Population - including only those participants who reported phonophobia at dose time.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 257 | 246 | 211
participants
  2 hrs post-dose | 11 | 25 | 15
  4 hrs post-dose | 15 | 57 | 24
  6 hrs post-dose | 21 | 49 | 30
  8 hrs post-dose | 21 | 57 | 30
  24 hrs post-dose | 33 | 79 | 61
  48 hrs post-dose | 34 | 71 | 52

11. Secondary Outcome: Number of Participants With Pain-freedom and Relief of Vomiting at 2, 4, 6, 8, 24 and 48 Hours Post-dose
Description: The number of participants with no pain and relief of vomiting in those participants for whom vomiting was present at dose time. Participants using rescue medication were removed from the participants with relief group for all subsequent timed assessments, regardless of pain and associated symptom evaluations at the specified time point.
Time Frame: as for outcome 2
Population: ITT Population - including only those participants who reported vomiting at dose time.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 17 | 22 | 16
participants
  2 hrs post-dose | 1 | 0 | 0
  4 hrs post-dose | 1 | 1 | 0
  6 hrs post-dose | 1 | 2 | 1
  8 hrs post-dose | 0 | 1 | 1
  24 hrs post-dose | 3 | 3 | 3
  48 hrs post-dose | 3 | 2 | 2

12. Secondary Outcome: Number of Participants With Relief From Sinus/Facial Pain at 2, 4, 6, 8, 24 and 48 Hours After Dosing in Those Who Also Had the Symptom at Dosing
Description: The number of participants with no pain and relief of sinus/facial pain in those participants for whom sinus/facial pain was present at dose time. Participants using rescue medication were removed from the participants with relief group for all subsequent timed assessments, regardless of pain and associated symptom evaluations at the specified time point.
Time Frame: as for outcome 2
Population: ITT Population - including only those participants who reported sinus/facial pain at dose time.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 133 | 148 | 134
participants
  2 hrs post-dose | 5 | 14 | 9
  4 hrs post-dose | 4 | 35 | 17
  6 hrs post-dose | 10 | 29 | 15
  8 hrs post-dose | 8 | 28 | 16
  24 hrs post-dose | 13 | 38 | 30
  48 hrs post-dose | 15 | 40 | 24

13. Secondary Outcome: Number of Participants With Relief From Neck Pain at 2, 4, 6, 8, 24 and 48 Hours After Dosing Who Also Had the Symptom at Baseline
Description: The number of participants with no pain and relief of neck pain in those participants for whom neck pain was present at dose time. Participants using rescue medication were removed from the participants with relief group for all subsequent timed assessments, regardless of pain and associated symptom evaluations at the specified time point.
Time Frame: as for outcome 2
Population: ITT Population - including only those participants who reported neck pain at dose time.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 194 | 181 | 188
participants
  2 hrs post-dose | 4 | 19 | 14
  4 hrs post-dose | 7 | 43 | 22
  6 hrs post-dose | 12 | 39 | 19
  8 hrs post-dose | 16 | 38 | 29
  24 hrs post-dose | 20 | 51 | 44
  48 hrs post-dose | 26 | 46 | 37

14. Secondary Outcome: Number of Participants With Pain Relief at 2, 4, 6, 8, 24 and 48 Hours After Dosing Moderate or Severe Baseline Pain
Description: Pain relief is defined as having no or mild pain and no use of rescue medication after dosing in those participants who had moderate or severe pain at dosing.
Time Frame: as for outcome 2
Population: ITT Population - only participants who reported moderate or severe baseline pain were included in this analysis.
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 309 | 307 | 296
participants
  2 hours post-dose | 76 | 148 | 114
  4 hours post-dose | 51 | 124 | 90
  6 hours post-dose | 48 | 107 | 66
  8 hours post-dose | 46 | 97 | 61
  24 hours post-dose | 62 | 127 | 88
  48 hours post-dose | 54 | 99 | 71

15. Secondary Outcome: Number of Participants Who Reported a Complete Symptom-Free Response at 2, 4, 6, 8, 24 and 48 Hours After Dosing
Description: Complete symptom-free is defined as migraine-free, neck pain-free, and sinus pain-free without the use of any rescue medication prior to the defined time point.
Time Frame: as for outcome 2
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 320 | 317 | 304
participants
  2 hours | 13 | 29 | 21
  4 hours | 19 | 68 | 36
  6 hours | 27 | 67 | 38
  8 hours | 29 | 68 | 38
  24 hours | 43 | 95 | 74
  48 hours | 47 | 86 | 62

16. Secondary Outcome: Mean Performance Index (PI) Scores at Time of Dosing and at 2, 4, 6, 8, 24 and 48 Hours After Dosing
Description: Overall cognition was assessed with a composite score (range 0-9) called the Performance Index, as derived from the number of correct responses per minute on subtests of the Mental Efficiency Workload Test (MEWT) cognitive battery. For a particular participant, lower scores indicate a negative impact, or worsened, general cognition; higher scores indicate improved cognition.
Time Frame: At time of dosing, and at 2, 4, 6, 8, 24, and 48 hours post-dose for each attack treated with study medication. All 3 migraine attacks were to have been treated within 19 weeks of randomization (when study medication was dispensed).
Population: ITT Population
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 320 | 317 | 304
scores on a scale
  Dose time | 7.36 (1.598) | 7.29 (1.534) | 7.30 (1.556)
  2 hours | 7.33 (1.606) | 7.37 (1.568) | 7.27 (1.579)
  4 hours | 7.44 (1.568) | 7.50 (1.576) | 7.38 (1.601)
  6 hours | 7.38 (1.658) | 7.43 (1.532) | 7.34 (1.482)
  8 hours | 7.45 (1.666) | 7.33 (1.632) | 7.33 (1.538)
  24 hours | 7.66 (1.524) | 7.82 (1.525) | 7.61 (1.494)
  48 hours | 7.78 (1.636) | 7.88 (1.351) | 7.69 (1.463)

17. Secondary Outcome: Mean Stanford Sleepiness (SS) Scale Scores at Time of Dosing and at 2, 4, 6, 8, 24 and 48 Hours After Dosing
Description: Participant alertness was evaluated with the 7-point modified SS scale, where 1 is "feeling active, vital, alert, wide awake", 2 is "still functioning at high levels, but not peak; able to concentrate", 3 is "awake, but relaxed; responsive but not fully alert", 4 is "somewhat foggy, let down", 5 is "foggy, losing interest in remaining awake", 6 is "sleepy, woozy, fighting sleep, prefer to lie down", and 7 is "no longer fighting sleep, sleep onset soon, having dream like thoughts".
Time Frame: Dose time, 2, 4, 6, 8, 24 and 48 hours post-dose. All 3 migraine attacks were to have been treated within 19 weeks of randomization (when study medication was dispensed).
Population: ITT Population. Only participants who responded to the SS scale at a particular time point were included in the analysis for that time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 318 | 316 | 304
units on a scale
  Dose time, n=318, 316, 304 | 3.94 (1.185) | 3.97 (1.156) | 4.00 (1.121)
  2 hours, n=275, 268, 251 | 3.88 (1.318) | 3.87 (1.481) | 3.88 (1.337)
  4 hours, n=249, 240, 234 | 3.75 (1.488) | 3.67 (1.718) | 3.91 (1.555)
  6 hours, n=215, 219, 210 | 3.78 (1.810) | 3.75 (1.870) | 3.82 (1.578)
  8 hours, n=195, 195, 186 | 3.85 (1.873) | 3.81 (2.061) | 3.91 (1.882)
  24 hours, n=252, 258, 241 | 2.73 (1.452) | 2.80 (1.516) | 2.78 (1.570)
  48 hours, n=215, 240, 218 | 2.56 (1.445) | 2.72 (1.453) | 2.60 (1.522)

18. Secondary Outcome: Efficacy Subscore as Measured by the Revised Patient Perception of Migraine (PPMQ-R) Questionnaire 24 Hours After Treating a Migraine
Description: The PPMQ-R questionnaire was used to assess participant satisfaction with migraine medication; the answers are used to generate a total score and 4 subscales scores for efficacy, functionality, ease-of-use and bothersomeness-of-side effects. The total score was calculated as the average of the efficacy, functionality and ease-of-use subscores. Subscores could range from 0 to 100; higher scores indicate greater satisfaction.
Time Frame: At 24 hours after dosing for each attack treated with study medication. All 3 migraine attacks were to have been treated within 19 weeks of randomization (when study medication was dispensed).
Population: ITT Population: those participants who provided any information for the PPMQ-R.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 224 | 254 | 234
scores on a scale | 55 (1.8) | 62 (1.7) | 56 (1.8)

19. Secondary Outcome: Functionality Subscore as Measured by the Revised Patient Perception of Migraine (PPMQ-R) Questionnaire 24 Hours After Taking Study Medication
Description: as for outcome 18
Time Frame: as for outcome 18
Population: ITT Population: those participants who provided any information for the PPMQ-R.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 224 | 254 | 234
scores on a scale | 55 (1.9) | 61 (1.8) | 56 (1.9)

20. Secondary Outcome: Ease-of-Use Subscore as Measured by the Revised Patient Perception of Migraine (PPMQ-R) Questionnaire 24 Hours After Taking Study Medication
Description: as for outcome 18
Time Frame: as for outcome 18
Population: ITT Population: those participants who provided any information for the PPMQ-R.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 224 | 254 | 234
scores on a scale | 79 (1.3) | 82 (1.3) | 78 (1.3)

21. Secondary Outcome: Bothersomeness-of-side Effect Subscore as Measured by the Revised Patient Perception of Migraine (PPMQ-R) Questionnaire 24 Hours After Taking Study Medication
Description: as for outcome 18
Time Frame: as for outcome 18
Population: ITT Population: those participants who provided any information for the PPMQ-R.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 224 | 254 | 234
scores on a scale | 88 (0.8) | 86 (0.8) | 89 (0.9)

22. Secondary Outcome: Total PPMQ-R Score as Measured With the Revised Patient Perception of Migraine (PPMQ-R) Questionnaire 24 Hours After Taking Study Medication
Description: as for outcome 18
Time Frame: as for outcome 18
Population: ITT Population: those participants who provided any information for the PPMQ-R.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 224 | 254 | 234
scores on a scale | 63 (1.5) | 68 (1.4) | 63 (1.5)

23. Secondary Outcome: Numbers of Participants Able to "Engage in Normal Activities Not Impaired" at Time of Dosing and 2, 4, 6, and 8 Hours After Dosing as Assessed by the CDQ (Clinical Disability Questionnaire)
Description: Clinical disability for each participant was assessed using the CDQ. This scale uses one question to assess ability to perform normal or usual activities. Responses are recorded on a 5-point scale, where 1 is "normal/not impaired", 2 is "mildly impaired", 3 is "moderately impaired", 4 is "severely impaired", and 5 is '"required bedrest".
Time Frame: At dosing and at 2, 4, 6 and 8 hours after dosing of each attack treated with study medication. All 3 migraine attacks were to have been treated within 19 weeks of randomization (when study medication was dispensed).
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Number analyzed (Participants) | 320 | 317 | 304
participants
  At dose time | 9 | 8 | 10
  2 hours | 19 | 33 | 29
  4 hours | 59 | 62 | 50
  6 hours | 76 | 77 | 60
  8 hours | 77 | 83 | 60

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time of first dose of study medication until the final study visit (within 19 weeks of randomization). Serious AEs were also collected if they occurred prior to dosing and were related to screening procedures.
Description: AEs and SAEs were assessed in the Safety Population (SP), comprised of all 442 participants treated at least once with study medication. Only a portion of the participants who were randomized comprise the SP. Reflecting the study's cross over design, AEs are categorized by the initial blinded treatment for the attack treated preceding AE onset.
Groups:
- Placebo: Participants who reported an SAE anytime after initial treatment with blinded placebo, but before another initial treatment with any other investigational product
- Treximet: Participants who reported an SAE anytime after initial treatment with blinded Treximet, but before another initial treatment with any other investigational product
- Butalbital-containing Combination Medication: Participants who reported an SAE anytime after initial treatment with blinded Butalbital-containing combination medication, but before another initial treatment with any other investigational product
Arm/Group | Placebo | Treximet | Butalbital-containing Combination Medication
Serious Adverse Events (participants affected / at risk) | 1/405 | 2/406 | 0/392
Other Adverse Events (participants affected / at risk) | 8/405 | 8/406 | 2/392
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=405) | Treximet (N=406) | Butalbital-containing Combination Medication (N=392)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=405) | Treximet (N=406) | Butalbital-containing Combination Medication (N=392)
Nausea (Gastrointestinal disorders) | 8 | 8 | 2

LIMITATIONS AND CAVEATS:
Enrolled participants included all those entering the screening part of the study. Randomized participants included only those who completed screening and completed the 2-week butalbital wash-out, and were successfully randomized to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.